CLINICAL TRIAL: NCT04144192
Title: Phase 1, Randomized, Comparative Pharmacokinetic Study of Bolus Intravenous Lidocaine 0.7 mg/kg, Lidocaine Patch 1.8%, and Lidocaine Patch 5% (Lidoderm®) in Healthy Subjects
Brief Title: Pharmacokinetic Study of Lidocaine Patch 1.8% Lidocaine Patch 5% (Lidoderm®) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scilex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SCI-LIDO-PK-001
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Healthy
MeSH Terms: interventions — Lidocaine; Transdermal Patch; Lidoderm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lidocaine Patch (Sequence AB) (Experimental): Subjects received all study treatments: a bolus IV injection of 0.7 mg/kg lidocaine IV in the morning of study Day 1, and then lidocaine patch treatment on Day 8 and Day 15. The sequence in which they received patch treatment was determined by random assignment. For subjects in Arm 1, 3 lidocaine 1.8% patches were applied on Day 8 and 3 Lidoderm® 5% patches were applied on Day 15.
  Interventions: Drug: Lidocaine patch 1.8%; Drug: Lidocaine 5% patch; Drug: Lidocaine 2% Injectable Solution
- Lidocaine Patch (Sequence BA) (Experimental): Subjects received all study treatments: a bolus IV injection of 0.7 mg/kg lidocaine IV in the morning of study Day 1, and then lidocaine patch treatment on Day 8 and Day 15. The sequence in which they received patch treatment was determined by random assignment. For subjects in Arm 2, 3 Lidoderm® 5% patches were applied on Day 8 and 3 lidocaine 1.8% patches were applied on Day 15.
  Interventions: Drug: Lidocaine patch 1.8%; Drug: Lidocaine 5% patch; Drug: Lidocaine 2% Injectable Solution

INTERVENTIONS:
Drug: Lidocaine patch 1.8%
  Other Names: Lidocaine topical system 1.8%
Drug: Lidocaine 5% patch
  Other Names: Lidoderm
Drug: Lidocaine 2% Injectable Solution

SUMMARY:
The purpose of this study is to characterize the comparative single-dose pharmacokinetics (bioequivalence) of lidocaine patch 1.8% (investigational product) versus Lidoderm® (lidocaine patch 5%,reference product).

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy based on by medical history, laboratory work, and physical exam
* Be at least 18 years of age to 65 years of age
* If childbearing potential, use of acceptable form of birth control
* In the case of females of childbearing potential, have a negative serum pregnancy test

Exclusion Criteria:

* Use of a prescription medication within 14 days or over-the-counter products within 7 days prior to administration of study medication
* Known hypersensitivity or allergy to any of the components of the lidocaine topical system formulation
* Any serious illness in the 4 weeks preceding the beginning of treatment that resulted in missed work or hospitalization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-04-28 (Actual); Primary Completion 2014-07-24 (Actual); Study Completion 2014-07-24 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of lidocaine | 0, 2, 4, 6, 9, 10, 11, 12, 13, 14, 16, 18, 20, 22, 24, 48 hours post-dose
  Peak plasma concentration of lidocaine after application of 3 patches for 12 hours
Area under the Plasma Concentration-Time Curve (AUC) from Time 0 to Time 48 hours | 0, 2, 4, 6, 9, 10, 11, 12, 13, 14, 16, 18, 20, 22, 24, 48 hours post-dose
  Area under the plasma concentration versus time curve from 0 to 48 hours of lidocaine in plasma
Area under the Plasma Concentration-Time Curve (AUC) from Time 0 to Time Infinity | 0, 2, 4, 6, 9, 10, 11, 12, 13, 14, 16, 18, 20, 22, 24, 48 hours post-dose
  Area under the plasma concentration versus time curve from 0 to infinite time of lidocaine in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Phillip LaStella, MD, Principal Investigator — TKL Research, Inc.

REFERENCES:
- [Derived] Gudin J, Argoff C, Fudin J, Greuber E, Vought K, Patel K, Nalamachu S. A Randomized, Open-Label, Bioequivalence Study of Lidocaine Topical System 1.8% and Lidocaine Patch 5% in Healthy Subjects. J Pain Res. 2020 Jun 22;13:1485-1496. doi: 10.2147/JPR.S237934. eCollection 2020. PMID 32606914